CLINICAL TRIAL: NCT04130802
Title: A Randomized, Double-masked, Vehicle-controlled Study Evaluating the Efficacy and Safety of Two Doses of OCS 01 Compared to Vehicle in the Treatment of Inflammation and Pain Following Cataract Surgery
Brief Title: OCS-01 in Treating Inflammation and Pain in Post-cataract Patients
Acronym: SKYGGN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oculis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DX-216
Record Dates: First submitted 2019-10-16; First posted 2019-10-17 (Actual); Results first posted 2022-03-15 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Inflammation Corneal; Pain, Postoperative
Keywords: post-cataract,; inflammation; Pain; post-surgery; corticosteroid; anterior chamber cells; flares
MeSH Terms: conditions — Keratitis; Pain, Postoperative; Inflammation; Pain

STUDY DESIGN:
Intervention Model Description: Randomized, double-masked, placebo (vehicle)-controlled study evaluating the efficacy and safety of two doses of OCS-01 compared to vehicle
Who Masked: Participant, Outcomes Assessor
Masking Description: For masking purposes, each dosing box and the pouches within it will be labeled either "AM" or "PM." Dosing boxes and pouches will be labeled this way regardless of whether the product within the 2 boxes is the same (i.e. OCS-01 BID and placebo treatment arms) or different (i.e. OCS-01 QD).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OCS-01 1.5% mg/mL QD (Experimental): eye drops
  Interventions: Drug: OCS-01 - Dexamethasone Cyclodextrin Nanoparticle Ophthalmic Suspension 1.5% mg/mL; Drug: Placebo
- OCS-01 1.5% mg/mL BID (Experimental): eye drops
  Interventions: Drug: OCS-01 - Dexamethasone Cyclodextrin Nanoparticle Ophthalmic Suspension 1.5% mg/mL
- Placebo (Vehicle) BID (Placebo Comparator): eye drops
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OCS-01 - Dexamethasone Cyclodextrin Nanoparticle Ophthalmic Suspension 1.5% mg/mL — OCS-01 eye drops
  Other Names: DexNP
  Arms: OCS-01 1.5% mg/mL BID; OCS-01 1.5% mg/mL QD
Drug: Placebo — Vehicle eye drops
  Other Names: Vehicle
  Arms: OCS-01 1.5% mg/mL QD; Placebo (Vehicle) BID

SUMMARY:
The DX-216 trial is a randomized, double-masked, placebo (vehicle)-controlled study evaluating the efficacy and safety of two doses of OCS-01 compared to vehicle in the treatment of inflammation and pain following cataract surgery. The primary objective is to evaluate the efficacy and safety of OCS-01 compared to placebo and the secondary objective is to evaluate the optimal dosing frequency (once a day [QD] or twice a day [BID]).

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-masked, placebo (vehicle)-controlled study, designed to evaluate the efficacy and safety of OCS-01 ophthalmic suspension (QD versus BID) compared to placebo in treating inflammation and pain following cataract surgery. Subjects will be randomized 1:1:1 to receive OCS-01 QD, OCS-01 BID, or placebo BID. Subjects will dose 1 drop in the study eye BID for 14 days, beginning 1 day post-surgery in the operated eye. The study will last up to 24 days, including a follow-up visit at Visit 7 (Day 22 ± 2).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent, approved by the appropriate ethics committee;
2. Be able to comply with the study requirements and visit schedule;
3. Be at least 18 years of age of either sex or any race;
4. Be planning to undergo unilateral cataract extraction via phacoemulsification and PCIOL implantation in the study eye;
5. Have an anterior chamber cell score ≥ 2 at Visit 2 (Day 1 [18 to 30 hours post-uncomplicated cataract surgery without vitreous loss]);
6. Have a pin-hole visual acuity (VA) without any other correction > 20 letters (approximately 20/400) in the operative eye and > 35 letters (approximately 20/200) in the fellow eye as measured using an Early Treatment for Diabetic Retinopathy Study (ETDRS) chart at Visit 1 (Day -1 to Day -28 [prior to surgery]);
7. Have a negative urine pregnancy test at Visit 1 (Day -1 to Day -28 [prior to surgery]),

Exclusion Criteria:

1. Have a known sensitivity or allergy to dexamethasone, corticosteroids, or any of the study medication's components;
2. Be monocular;
3. Have any intraocular inflammation (e.g. white blood cells or flare) present in either eye at the Visit 1 (Day -1 to Day -28 [prior to surgery]) slit lamp examination;
4. Have a score > 0 on the Ocular Pain Assessment at Visit 1 (Day -1 to Day -28 [prior to surgery]) in the study eye;
5. Use anti-inflammatory agents, analgesics/pain relievers (including opioids, narcotics, and other pain medications), or immunomodulating agents, systemically or in either eye, and/or use medications for benign prostatic hyperplasia (BPH), from the washout period through the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Medical cennre, Petaluma, California
  - Medical center, Roseburg, Oregon
  - Medical center, Houston, Texas
  - Medical center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohira A, Hara K, Johannesson G, Tanito M, Asgrimsdottir GM, Lund SH, Loftsson T, Stefansson E. Topical dexamethasone gamma-cyclodextrin nanoparticle eye drops increase visual acuity and decrease macular thickness in diabetic macular oedema. Acta Ophthalmol. 2015 Nov;93(7):610-5. doi: 10.1111/aos.12803. Epub 2015 Jul 23. PMID 26201996
- [Background] Tanito M, Hara K, Takai Y, Matsuoka Y, Nishimura N, Jansook P, Loftsson T, Stefansson E, Ohira A. Topical dexamethasone-cyclodextrin microparticle eye drops for diabetic macular edema. Invest Ophthalmol Vis Sci. 2011 Oct 10;52(11):7944-8. doi: 10.1167/iovs.11-8178. PMID 21896859
- [Background] Johannesson G, Moya-Ortega MD, Asgrimsdottir GM, Lund SH, Thorsteinsdottir M, Loftsson T, Stefansson E. Kinetics of gamma-cyclodextrin nanoparticle suspension eye drops in tear fluid. Acta Ophthalmol. 2014 Sep;92(6):550-6. doi: 10.1111/aos.12334. Epub 2013 Dec 24. PMID 24373641
- [Background] Saari KM, Nelimarkka L, Ahola V, Loftsson T, Stefansson E. Comparison of topical 0.7% dexamethasone-cyclodextrin with 0.1% dexamethasone sodium phosphate for postcataract inflammation. Graefes Arch Clin Exp Ophthalmol. 2006 May;244(5):620-6. doi: 10.1007/s00417-005-0124-2. Epub 2005 Oct 11. PMID 16217662
- [Derived] Korenfeld M, Gira J, Jong K, Martel J, Vold S, Walters T, Usner D, Donnenfeld E. OCS-01 (Novel Topical Dexamethasone Formulation) in Inflammation and Pain Post Cataract Surgery: A Randomized, Double-Masked, Vehicle-Controlled Study. Clin Ther. 2022 Dec;44(12):1577-1587. doi: 10.1016/j.clinthera.2022.11.003. Epub 2022 Dec 8. PMID 36503736

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OCS-01 1.5% mg/mL QD | OCS-01 1.5% mg/mL BID | Placebo (Vehicle) BID
Started | 51 | 51 | 51
Completed | 50 | 50 | 48
Not Completed | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OCS-01 1.5% mg/mL QD | OCS-01 1.5% mg/mL BID | Placebo (Vehicle) BID | Total
Number analyzed (Participants) | 51 | 51 | 51 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 22 | 15 | 50
  >=65 years | 38 | 29 | 36 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (6.86) | 65.8 (6.59) | 67.5 (8.41) | 67.1 (7.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 36 | 32 | 101
  Male | 18 | 15 | 19 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 3 | 8 | 4 | 15
  White | 47 | 42 | 47 | 136
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 51 | 51 | 51 | 153

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Absence of Anterior Chamber Cells (i.e. Score of '0')
Description: Absence of anterior chamber cells as measured by slit beam with fluorescein. The anterior chamber cell count was recorded as the actual number of cells observed if ≤10 cells were seen, otherwise a range was reported. The observed anterior chamber cell count at Visit 6 was used and categorized for analysis as follows:
  * Absence of anterior chamber cells: anterior chamber cell count of 0 / Grade 0
  * Presence of anterior chamber cells: anterior chamber cell count of 1 or more / Grade 1, 2, 3, or 4
Time Frame: at Day 15 (visit 6)
Measure: Number; unit: participants
Arm/Group | OCS-01 1.5% mg/mL QD | OCS-01 1.5% mg/mL BID | Placebo (Vehicle) BID
Number analyzed (Participants) | 51 | 51 | 51
participants | 26 | 34 | 10

2. Primary Outcome: Number of Subjects With Absence of Ocular Pain (i.e. Score of '0')
Description: Absence of pain as assessed by Ocular Pain Grading Scale (Min 0, Max 10) in which 0 is no pain and 10 is the worst possible. Ocular pain was assessed by the patient at screening and at each follow-up visit, utilizing a numerical pain rating scale. Scores ranged from 0 to 10, where 0 = No Pain and 10 = Severe Pain, such that larger scores corresponded to higher levels of pain.
Time Frame: at Day 4 (visit 4)
Measure: Number; unit: participants
Arm/Group | OCS-01 1.5% mg/mL QD | OCS-01 1.5% mg/mL BID | Placebo (Vehicle) BID
Number analyzed (Participants) | 51 | 51 | 51
participants | 37 | 32 | 23

ADVERSE EVENTS:
Time Frame: The AEs were queried at visit 2 (Day 1, 18 - 30h post surgery), visit 4 (Day 4) , visit 5 (Day 8), visit 6 (Day 15) & visit 7 (Day 22)
Arm/Group | OCS-01 1.5% mg/mL QD | OCS-01 1.5% mg/mL BID | Placebo (Vehicle) BID
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51 | 1/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 1/51 | 1/51
Other Adverse Events (participants affected / at risk) | 17/51 | 10/51 | 20/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OCS-01 1.5% mg/mL QD (N=51) | OCS-01 1.5% mg/mL BID (N=51) | Placebo (Vehicle) BID (N=51)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) — TEAE serious, severe, not suspected related to study drug. Outcome of this event was fatal
noninfectious endophthamitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — TEAE serious, severe, unexpected and suspected of related to study drug (SUSAR) Classified as recovering/resolving
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — reported prior to study drug administration. Was considered serious, severe, and nos suspected of being related to study drug. Outcome was classified as resolved/recovered
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OCS-01 1.5% mg/mL QD (N=51) | OCS-01 1.5% mg/mL BID (N=51) | Placebo (Vehicle) BID (N=51)
conjunctival hyperaemia (Eye disorders) | 3 (3) | 2 (2) | 8 (8)
corneal edema (Eye disorders) | 5 (5) | 1 (1) | 8 (8)
anteror chamber inflammation (Eye disorders) | 1 (1) | 3 (3) | 0 (0)
iritis (Eye disorders) | 3 (3) | 0 (0) | 2 (2)
vitreous detachment (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
foreign body sensation in eyes (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
posterior capsule opacification (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
anterior chamber flare (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
ciliary hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
conjunctival oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
corneal disorder (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
eye inflammation (Eye disorders) | 1 (1) | 0 (0) | 2 (2)
keratic precipitates (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
lacrimination increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
macular oedema (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
non infectious endophtalmitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
retinal haemmorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
retinal pigment epitheliopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
anterior chamber cell (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
eye pain (Eye disorders) | 0 (0) | 0 (0) | 4 (4)
photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
photopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
punctate keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
pupillary disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Instillation site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
instillation site foreign body sensation (General disorders) | 0 (0) | 0 (0) | 1 (1)
intraocular pressure increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Dandruff (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
vitreous detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agrees not to publish/present the results until such time as the aggregate study results are published. After such time, Investigator may publish the results in accordance with the following: Investigator shall submit to Sponsor any such proposed publication/presentation resulting from or relating to the Study at least 60 days prior to the submission for publication. Sponsor may require the delay of publication/presentation for an additional period of time not to exceed 120 days.

DOCUMENTS (2):
  • Study Protocol (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT04130802/Prot_002.pdf
  • Statistical Analysis Plan (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT04130802/SAP_003.pdf